CLINICAL TRIAL: NCT03593902
Title: Autologous Hematopoietic Stem Cell Transplant for Patients With Systemic Sclerosis and Cardiac Dysfunction
Brief Title: Cardiac Safe Transplants for Systemic Sclerosis
Acronym: CAST
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI Sabbatical
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAD.CAST.2018
Record Dates: First submitted 2018-06-28; First posted 2018-07-20 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-06

CONDITIONS: Systemic Sclerosis; Scleroderma
Keywords: Autologous Stem Cell Transplantation; Hematopoietic Stem Cell Transplant
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Rituximab; fludarabine; fludarabine phosphate; Cyclophosphamide; Mesna; thymoglobulin; Antilymphocyte Serum; Methylprednisolone; Methylprednisolone Hemisuccinate; Methylprednisolone Acetate; Granulocyte Colony-Stimulating Factor; Filgrastim; Immunoglobulins, Intravenous; Octagam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Experimental): Hematopoietic Stem Cell Therapy will be performed as follows: Autologous stem cells will be infused after conditioning with rituximab, fludarabine, cyclophosphamide, Mesna, rATG (rabbit), and methylprednisolone. Granulocyte-colony stimulating factor (G-CSF) and intravenous immunoglobulin (IVIg) will be administered post-transplant.
  Interventions: Drug: Rituximab; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mesna; Drug: rATG; Drug: Methylprednisolone; Drug: G-CSF; Biological: IVIg; Biological: Autologous Stem Cells

INTERVENTIONS:
Drug: Rituximab — Monoclonal antibody therapy used to treat certain autoimmune diseases and types of cancer
  Other Names: Rituxan
Drug: Fludarabine — A chemotherapy medication commonly used in the treatment of leukemia and lymphoma
  Other Names: Fludara
Drug: Cyclophosphamide — A medication used as chemotherapy and to suppress the immune system
  Other Names: Cytoxan
Drug: Mesna — A medication used in those taking cyclophosphamide or ifosfamide to decrease the risk of bleeding from the bladder
  Other Names: Mesnex
Drug: rATG — A rabbit polyclonal antibody to lymphocytes
  Other Names: Thymoglobulin; Anti-Thymocyte Globulin (Rabbit)
Drug: Methylprednisolone — A corticosteroid medication used to suppress the immune system and decrease inflammation
  Other Names: Solu-Medrol; Depo-Medrol
Drug: G-CSF — A glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream
  Other Names: Neupogen; Filgrastim; Granix; Zarxio
Biological: IVIg — Pooled immunoglobulin (IgG) from thousands of plasma donors that has immunomodulatory and anti-inflammatory effects
  Other Names: Bivagam; Carimune NF; Gammagard; Privigen; Octagam
Biological: Autologous Stem Cells — Infusion of patient's own stem cells

SUMMARY:
This study is designed to treat systemic sclerosis (scleroderma) patients with an autologous stem cell transplant using a regimen of immune suppressant drugs and chemotherapy that is less toxic to your heart.

DETAILED DESCRIPTION:
The autologous hematopoietic stem cell transplant used in this research study is an investigational procedure that uses cyclophosphamide and fludarabine (chemotherapy), rabbit anti-thymocyte globulin (rATG) (a protein that kills the immune cells that are thought to be causing your disease), and rituximab (a biologic drug that targets B cells of your immune system). After use of these treatments, the patient will receive their own previously collected blood stem cells (autologous stem cell transplant). The ability of these experimental treatments to stop relapses and progression (worsening) of your systemic sclerosis will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 65 years old at the time of pre-transplant evaluation
2. An established diagnosis of systemic sclerosis
3. Diffuse cutaneous systemic sclerosis with involvement proximal to the elbow or knee and a modified Rodnan Skin Score of ≥ 14 (see Appendix A)

AND

Any one of the following:

1. DLCO < 80% of predicted or decrease in lung function (DLCO, DLCO/VA or FVC) of 10% or more over 12 months.
2. Pulmonary fibrosis or alveolitis on CT scan or chest x-ray (ground glass appearance of alveolitis).
3. Abnormal EKG (non-specific ST-T wave abnormalities, low QRS voltage, or ventricular hypertrophy), or pericardial effusion or pericardial enhancement without constriction on MRI
4. Gastrointestinal tract involvement confirmed on radiological study. Radiologic findings of scleroderma are small bowel radiographs showing thickened folds with dilated loops, segmentation, and flocculation +/- diverticula, or pseudodiverticula. A hide-bound appearance may be present (e.g. dilated and crowded circular folds). GI involvement may also be confirmed by D-xylose malabsorption, patulous esophagus on high-resolution computed tomography (HRCT), or esophageal manometry.

OR

Limited cutaneous systemic sclerosis (SSc) (modified Rodnan Skin Score <14) with lung involvement defined as active alveolitis on bronchoalveolar lavage (BAL), ground-glass opacity on CT scan, a DLCO < 80% predicted, or decrease in lung function (DLCO/VA, DLCO, FVC) of 10% or more in last 12 months.

Other Inclusion Criteria for "CAST" Conditioning Regimen (presence of any of the following):

1. Septal flattening or D-sign on MRI (without deep breathing)
2. PASP >40 mm Hg or >45 mm Hg with fluid challenge*
3. mPAP >25 mm Hg or >30 mm Hg with fluid challenge*
4. Non-ischemia diffuse ventricular hypokinesis or non-ischemia wall hypokinesis

   * Fluid challenge is 1000 ml normal saline over 10 minutes. Fluid challenge will not be done if right atrial pressure is >13 mm Hg at rest or pulmonary capillary wedge pressure is >20 mm Hg at rest.

Exclusion Criteria:

1. Active ischemic heart disease or untreated coronary artery disease
2. Untreated life-threatening cardiac arrhythmia on EKG or 24-hour holter
3. Pericardial effusion > 1 cm on cardiac MRI unless successful pericardiocentesis has been performed
4. LVEF <35%
5. End-stage lung disease characterized by TLC<45% of predicted value, or DLCO hemoglobin corrected < 30 % predicted.
6. Creatinine clearance <40 by 24-hour urine
7. History of breast implants that have not been removed (unless they cannot be surgically removed due to risks of surgery)
8. Liver cirrhosis, transaminases >2x of normal limits, or bilirubin > 2.0 unless due to Gilbert's disease
9. Uncontrolled diabetes mellitus or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment
10. Prior history of malignancy
11. Positive pregnancy test, inability or unable to pursue effective means of birth control, or failure to willingly accept or comprehend irreversible sterility as a side effect of therapy
12. Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
13. Major hematological abnormalities such as platelet count < 100,000/ul or absolute neutrophil count (ANC) < 1000/ul
14. HIV positive
15. Hepatitis B or C positive
16. PASP >50 mmHg without fluid challenge
17. mPAP >34 mmHg without fluid challenge
18. Coronary artery disease not reversed by cardiology and interventional radiology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burt RK, Han X, Quigley K, Arnautovic I, Shah SJ, Lee DC, Freed BH, Jovanovic B, Helenowski IB. Cardiac safe hematopoietic stem cell transplantation for systemic sclerosis with poor cardiac function: a pilot safety study that decreases neutropenic interval to 5 days. Bone Marrow Transplant. 2021 Jan;56(1):50-59. doi: 10.1038/s41409-020-0978-2. Epub 2020 Jul 1. PMID 32612255

RESULTS

PARTICIPANT FLOW:
Groups:
- Hematopoietic Stem Cell Transplantation: Hematopoietic Stem Cell Therapy will be performed as follows: Autologous stem cells will be infused after conditioning with rituximab, fludarabine, cyclophosphamide, Mesna, rATG (rabbit), and methylprednisolone. Granulocyte-colony stimulating factor (G-CSF) and intravenous immunoglobulin (IVIg) will be administered post-transplant.
  Rituximab: Monoclonal antibody therapy used to treat certain autoimmune diseases and types of cancer
  Fludarabine: A chemotherapy medication commonly used in the treatment of leukemia and lymphoma
  Cyclophosphamide: A medication used as chemotherapy and to suppress the immune system
  Mesna: A medication used in those taking cyclophosphamide or ifosfamide to decrease the risk of bleeding from the bladder
  rATG: A rabbit polyclonal antibody to lymphocytes
  Methylprednisolone: A corticosteroid medication used to suppress the immune system and decrease inflammation
  G-CSF: A glycoprotein that stimulates the bone marrow to produce granulocytes and
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hematopoietic Stem Cell Transplantation: Hematopoietic Stem Cell Therapy will be performed: Autologous stem cells will be infused after conditioning with rituximab, fludarabine, cyclophosphamide, Mesna, rATG (rabbit), and methylprednisolone. Granulocyte-colony stimulating factor (G-CSF) and intravenous immunoglobulin (IVIg) will be administered post-transplant.
  Rituximab: Monoclonal antibody therapy used to treat certain autoimmune diseases and types of cancer
  Fludarabine: A chemotherapy medication commonly used in the treatment of leukemia and lymphoma
  Cyclophosphamide: A medication used as chemotherapy and to suppress the immune system
  Mesna: A medication used in those taking cyclophosphamide or ifosfamide to decrease the risk of bleeding from the bladder
  rATG: A rabbit polyclonal antibody to lymphocytes
  Methylprednisolone: A corticosteroid medication used to suppress the immune system and decrease inflammation
  G-CSF: A glycoprotein that stimulates the bone marrow to produce granulocytes and
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Modified Rodnan skin score [Mean (Full Range); unit: units on a scale] — The modified Rodnan skin score (MRSS) is a measure for skin disease in systemic scleroderma and is calculated by summation of skin thickness in 17 different body sites. The range is 0 (normal skin thickness to 51 (severe thickness).
  units on a scale | 25 [0 to 51]

OUTCOME MEASURES:

1. Primary Outcome: Change in Skin Score by mRSS
Description: Defined by at least a 25% improvement (decline) in skin score by modified Rodnan skin score (mRSS) if skin score is greater than 14 on enrollment. If skin score is less than 14 on enrollment, improvement is defined by at least a 5% improvement on mRSS. The modified Rodnan skin score (MRSS) is a measure for skin disease in scleroderma and is calculated by summation of skin thickness in 17 different body sites. The scale ranges from at total score of normal skin thickness (0) to severe thickness (51).
Time Frame: Pre Treatment and Post Treatment
Population: The number analyzed in one or more rows differs from the overall number analyzed because some patients did not follow up after the treatment.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 9
units on a scale
  Pre Treatment | 25 [4 to 48]
  Post Treatment: number analyzed (Participants) | 6
  Post Treatment | 16 [2 to 30]

2. Secondary Outcome: Survival of Treatment
Description: Survival of Hematopoietic Stem Cell Transplant during treatment and post treatment up to 1 year.
Time Frame: During Treatment and Post Treatment up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: During Treatment and the First 100 days Post Treatment
Description: Grade 4 Toxicities
Groups:
- Hematopoietic Stem Cell Transplantation: Hematopoietic Stem Cell Therapy will be performed as follows: Autologous stem cells will be infused after conditioning with rituximab, fludarabine, cyclophosphamide, Mesna, rATG (rabbit), and methylprednisolone. Granulocyte-colony stimulating factor (G-CSF) and intravenous immunoglobulin (IVIg) will be administered post-transplant.
  Rituximab: Monoclonal antibody therapy used to treat certain autoimmune diseases and types of cancer
  Fludarabine: A chemotherapy medication commonly used in the treatment of leukemia & lymphoma
  Cyclophosphamide: A medication used as chemotherapy and to suppress the immune system
  Mesna: A medication used in those taking cyclophosphamide or ifosfamide to decrease the risk of bleeding from the bladder
  rATG: A rabbit polyclonal antibody to lymphocytes
  Methylprednisolone: A corticosteroid medication used to suppress the immune system and decrease inflammation
  G-CSF: A glycoprotein that stimulates the bone marrow to produce granulocytes and
Arm/Group | Hematopoietic Stem Cell Transplantation
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Early termination of study due to PI Sabbatical led to small number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT03593902/SAP_000.pdf
  • Study Protocol (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT03593902/Prot_002.pdf